CLINICAL TRIAL: NCT06377813
Title: Effect of Combined Mode-Kinetic Chain Exercise With and Without Core Stability Exercises on Pain, Range of Motion, Quality of Life on Patients With Knee Osteoarthritis
Brief Title: Combined Mode-Kinetic Chain Exercise With and Without Core Stability Exercises on Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR& AHS/23/01100/Maryam
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: Kinematic Chain Exercises, Knee Osteoarthritis, Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group will include 24 participants, the interventions will be given for 35-45 mins. All the participants will follow the same standardized exercise protocol 5 days a week, for 12 weeks.
  Interventions: Other: Mode-Kinetic Chain Exercise With Core Stability Exercises
- Group B (Active Comparator): This group will also include 24 participants, the interventions will be given for 20-30 mins. All the participants will follow the same standardized exercise protocol 5 days a week, for 12 weeks.
  Interventions: Other: Mode-Kinetic Chain Exercise

INTERVENTIONS:
Other: Mode-Kinetic Chain Exercise With Core Stability Exercises — the interventions will be given for 35-45 mins. All the participants will follow the same standardized exercise protocol 5 days a week, for 12 weeks.
  Arms: Group A
Other: Mode-Kinetic Chain Exercise — the interventions will be given for 35-45 mins. All the participants will follow the same standardized exercise protocol 5 days a week, for 12 weeks.
  Arms: Group B

SUMMARY:
The goal of this [type of study: Randomized control trial] is to [ see the effects of Combined Mode Kinetic Chain Exercises along with or without core stability exercises on pain, range of motion and disability ] in [ in patients with Knee Osteoarthritis].The main question it aims to answer is:

Wether core stability exercises is effective if performed along with Combined chain kinetic exercises to improves the condition of Knee Osteoarthritis? Group A will receive Core Stability Exercises along with Combined Chain Kinetic Exercises and Group B will receive combined Chain Kinetic Exercises.

DETAILED DESCRIPTION:
Knee joint Osteoarthritis is a prevalent and multifaceted condition, affecting a substantial portion of the general population (roughly 13% of women and 10% of men 60 years). Different techniques and treatment methods have been used to treat knee osteoarthritis. In this study, I will be identifying that core stability exercise if performed along with Combined chain kinetic exercise brings benefits to the patients of knee osteoarthritis. One of the techniques is Combined Chain Kinetic Exercise that i will be applying on both groups. The other one is the set of Core stability exercises.

The research involves two intervention groups (Group A and Group B) receiving specific treatments over 60 sessions within an twelve-week period. Group A incorporates the Combined Chain Kinetic Exercise,Core stability exercises, and transcutaneous electrical nerve stimulation (TENS) with a heating pad. Group B undergoes hot packs and TENS, followed by Combined Chain Kinetic Exercise, encompassing pain levels, range of motion (ROM), and Knee Injury and Osteoarthritis Outcome Score (KOOS) scores, will be evaluated using the Numeric Pain Rating Scale, Goniometer, and KOOS. Data analysis will employ SPSS version 26. Data will be collected at baseline, immediately post-intervention, and at follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 70 years with Knee Osteoarthritis

Exclusion Criteria:

* Participants suffering from any other condition of knee joint or if they are in active infection state

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 12 weeks
  NPRS consists of a scale with 0-10 readings. The zero denotes no pain while 1, 2, 3 denotes to mild pain, 4, 5, 6 denotes to moderate pain while 7-10 denotes to severe pain.
Kellgren and Lawrence system for classification of Osteoarthritis | 12 Weeks
  This classification system consists of 5 grades with Grade 0 indicating normal joint and Grade 4 as maximal osteoarthritic activity in joint
Knee Injury and Osteoarthritic outcome score (KOOS) | 12 weeks
  The KOOS has five separate subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)
Goniometer | 12 weeks
  Active range of Motion of the patient will be assessed using a universal goniometer for knee joint flexion and extension. the data will be collected at baseline knee joint goniometry

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah, Lahore 54000
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No